CLINICAL TRIAL: NCT04977271
Title: Serotonin-Norepinephrine Reuptake Inhibitors for the Prevention and Treatment of Pain, Depression, and Anxiety in Patients With Head & Neck Cancer
Brief Title: Mood Disorders in Head and Neck Cancer Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: study never opened
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Harishanker Jeyarajan, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007057
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Depressive Disorder; Head and Neck Cancer
MeSH Terms: conditions — Depressive Disorder; Head and Neck Neoplasms | interventions — Venlafaxine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Starting dose of oral venlafaxine immediate release (IR) 37.5 mg BID, to be taken with food. The dosing will be increased at a rate of 75mg per week for 3 weeks, to reach a desired dose of 300mg per day, taken as 150mg BID.
  For patients with hepatic impairment, severe renal impairment, or end-stage kidney disease, the starting dose is 37.5 mg once daily, and the dose is increased by increments of 37.5 mg per day, to a maximum of 187.5 mg per day, taken as 93.75 mg BID.
  Interventions: Drug: Venlafaxine
- Control Group (No Intervention): No intervention will be provided for this group

INTERVENTIONS:
Drug: Venlafaxine — The Immediate Release generic formulation of this drug will be used due to its ability to be crushed for those patients who rely on parenteral administration of medications.
  Other Names: Effexor
  Arms: Treatment Group

SUMMARY:
The purpose of this research study is to initiate a pharmacotherapy protocol for at-risk patients with newly diagnosed head and neck cancer in order to decrease the incidence of anxiety, depression, and uncontrolled pain during cancer treatment.

DETAILED DESCRIPTION:
Patients requiring treatment of his or her newly diagnosed mucosal or cutaneous head and neck cancer per standard of care guidelines that meet all enrollment criteria will be identified and enrolled after obtaining informed consent. This will occur in the clinic setting, and subsequent screening and work up will be performed.

Enrolled patients will be randomized into one of the two study groups (Treatment v Control) via a computer-based program.

Treatment Group: Participants will be prescribed a starting dose of venlafaxine immediate release (IR) 37.5 mg twice daily. The IR formulation was selected due to its ability to be crushed for those patients who rely on parenteral administration of medications. The dosing will be increased at a rate of 75mg per week, to reach a desired dose of 300mg, divided into 150mg BID dosing. This dosing was selected due to the need for at least 150mg to see noradrenergic effects. For patients with hepatic impairment, severe renal impairment, or end-stage kidney disease, the starting dose is 37.5 mg once daily, and the dose is increased by increments of 37.5 mg per day, to a maximum of 187.5 mg per day, given in two divided doses.

Control Group: Participants will not receive any pharmacological treatment.

Patients in the Treatment Group will meet with a dedicated research collaborator via telephone on a weekly visit (for a maximum of 3 visits) as the medication is being titrated up to ensure tolerability. If at any point there are side effects or concerns regarding tolerability of medication, a collaborating psychiatrist who specializes in treatment of depression is available for consultation.

Patients in both groups will follow up 6-8 weeks after beginning their chosen treatment regimen for their HNC as determined for them by their standard of care evaluation. They will complete all of the study questionnaires at this visit. Vital signs will be collected at this visit as well as concomitant medications and any adverse events they may be experiencing.

Follow-up visits will continue every three months following this visit per the patient's standard of care return to clinic visits. It is anticipated that participants will be seen in clinic during Months 6, 9, and 12 as follow up for their standard of care treatment regimen. Vital signs, concomitant medications, adverse events, and responses to questionnaires will be collected at these visits.

Participant duration will be up to one year. If at any point, patients meet criteria for MDD, they will be referred to a mental health counselor.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 18 years or older
4. Ability to speak and understand English
5. Have a recently diagnosed cutaneous or mucosal malignancy
6. Scheduled to undergo treatment for their malignancy (surgical or nonsurgical) with curative intent
7. Ability to take medication (by mouth or via parenteral route)
8. Willing to adhere to the study drug's dosing protocol

Exclusion Criteria:

1. Age less than 18 years
2. Inability to speak or understand English
3. Primary malignancy of thyroid or parathyroid origin
4. Currently meet diagnostic criteria for psychosis, schizophrenia, or moderate/severe major depressive disorder (MDD)
5. Currently receiving medication as treatment for depression or anxiety
6. Known allergic reaction to components of study drug
7. Have uncontrolled pain or chronic pain disorder
8. Treatment with another investigational drug or other intervention within 30 days
9. Females of child-bearing age who are pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
The rate of depression in patients undergoing treatment for head and neck cancer (HNC) | Baseline to 12 months
  The degree of depression in patients who currently do not show signs of depression at the beginning of undergoing HNC treatment. This will be assessed using the following validated questionnaires: Patient-Health Questionnaire (PHQ-9) and the Quick Inventory of Depressive Symptomatology (QIDS SR-16). For both questionnaires, an increase in score is considered to show a higher degree of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Grayson, MD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/71/NCT04977271/Prot_000.pdf